CLINICAL TRIAL: NCT01815502
Title: Response to Sildenafil in Patients With Fontan Physiology, A Pressure-volume Loop Analysis
Brief Title: Study of Effects of Sildenafil on Patients With Fontan Heart Circulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVL Fontan; AHA (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Single Ventricle Heart Disease After Fontan Surgery
Keywords: Single ventricle; Fontan; Sildenafil; Pressure-Volume Loops
MeSH Terms: conditions — Univentricular Heart | interventions — Cardiac Catheterization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dobutamine + Sildenafil (Experimental): Sildenafil will be given an one time dose 30 to 90 minutes prior to cardiac catheterization. Sildenafil will be given at a dose 1 milligram per kilogram with a maximum of 20 milligrams. During the catheterization patients will have specialized catheter placed in the heart that measures pressure and volume simultaneously. The patients will undergo an infusion of dobutamine up to 10 micrograms per kilogram per minute to mimic exercise for up to ten minutes..
  Interventions: Diagnostic Test: Cardiac catheterization
- Dobutamine + placebo (Placebo Comparator): Patients will be given a one time dose of sugar pill 30 to 90 minutes prior to cardiac catheterization.During the catheterization patients will have specialized catheter placed in the heart that measures pressure and volume simultaneously. The patients will undergo an infusion of dobutamine up to 10 micrograms per kilogram per minute to mimic exercise for up to ten minutes..
  Interventions: Diagnostic Test: Cardiac catheterization

INTERVENTIONS:
Diagnostic Test: Cardiac catheterization — All patients will receive a dobutamine infusion during catheterization. Patients were 1:1 randomized to a single dose of 1 mg/kg of sildenafil (max dose of 20 mg) or placebo 30-90 min prior to beginning of catheterization.

SUMMARY:
The study will investigate the cardiovascular effects of sildenafil on patients with Fontan circulation. Recent studies suggest that sildenafil may improve exercise in patients with Fontan circulation. However, why this occurs is not known. The study will used specialized catheters to measure pressure and volume. The measure of pressure and volume leads to more detailed analysis of heart function. Patients will receive either sugar pill or sildenafil prior to catheterization. It is believed that sildenafil will improve relaxation and contraction of the heart.

DETAILED DESCRIPTION:
Modifications to surgical procedures and medical treatment have led to a rapidly declining mortality rates in patients with single-ventricle heart disease (SV). However, SV patients still suffer from lower quality of life, decreased exercise capacity, worse neurodevelopmental outcomes and many other morbidities. While patients with SV circulation only make a small portion of all congenital heart diseases, 2-4 %, they require a great deal of resource utilization.

Standard medical treatments for adult heart failure have not had the same success in the SV population. Phosphodiesterase 5 (PDE5) inhibitors have recently become a frequently used medication class in patients with SV heart disease to treat pulmonary hypertension, heart failure, as well as "Fontan" failure (i.e., plastic bronchitis and protein-losing enteropathy). While there have been findings of improved measures of exercise capacity and some reports of improved symptoms of heart failure, the physiologic mechanisms behind these findings are not completely understood. There have been reports, indicating that the phosphodiesterase five inhibitors improve ventricular function in biventricular circulation patients and animal models. The aim of our study was to investigate the effect of acute PDE5 inhibition on ventricular function in SV patients after the final palliative surgery, the Fontan procedure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a congenital heart defect that leads to single ventricle physiology
* Previously performed Fontan surgery

Exclusion Criteria:

* The use of phosphodiesterase type 5 (PDE5) inhibitors at the time of catheterization of within 1 month of catheterization

  * Unstable arrhythmia at the time of catheterization
  * History of unstable arrhythmia within 2 months of catheterization
  * Venous, arterial or cardiac malformation that precludes the proper placement of a microconductance catheter
  * Allergy to sildenafil or previous significant adverse reaction to sildenafil (e.g. hypotension)

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Butts, M.D., Principal Investigator — Medical University of South Carolina; Andrew M Atz, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Goldberg DJ, French B, McBride MG, Marino BS, Mirarchi N, Hanna BD, Wernovsky G, Paridon SM, Rychik J. Impact of oral sildenafil on exercise performance in children and young adults after the fontan operation: a randomized, double-blind, placebo-controlled, crossover trial. Circulation. 2011 Mar 22;123(11):1185-93. doi: 10.1161/CIRCULATIONAHA.110.981746. Epub 2011 Mar 7. PMID 21382896
- [Background] Goldberg DJ, French B, Szwast AL, McBride MG, Marino BS, Mirarchi N, Hanna BD, Wernovsky G, Paridon SM, Rychik J. Impact of sildenafil on echocardiographic indices of myocardial performance after the Fontan operation. Pediatr Cardiol. 2012 Jun;33(5):689-96. doi: 10.1007/s00246-012-0196-9. Epub 2012 Feb 14. PMID 22331056
- [Derived] Butts RJ, Chowdhury SM, Baker GH, Bandisode V, Savage AJ, Atz AM. Effect of Sildenafil on Pressure-Volume Loop Measures of Ventricular Function in Fontan Patients. Pediatr Cardiol. 2016 Jan;37(1):184-91. doi: 10.1007/s00246-015-1262-x. Epub 2015 Sep 26. PMID 26409473

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Sildenafil will be given an one time dose 30 to 90 minutes prior to catheterization. Sildenafil will be given at a dose 1 milligram per kilogram with a maximum of 20 milligrams. During the catheterization patients will have specialized catheter placed in the heart that measures pressure and volume simultaneously. The patients will undergo an infusion of dobutamine up to 10 micrograms per kilogram per minute to mimic exercise for up to ten minutes..
  Dobutamine: Patients will receive a dobutamine infusion during catheterization.
- Sugar Pill: Patients will be given a one time dose of sugar pill 30 to 90 minutes prior to catheterization.During the catheterization patients will have specialized catheter placed in the heart that measures pressure and volume simultaneously. The patients will undergo an infusion of dobutamine up to 10 micrograms per kilogram per minute to mimic exercise for up to ten minutes..
  Dobutamine: Patients will receive a dobutamine infusion during catheterization.
Period: Overall Study
Arm/Group | Sildenafil | Sugar Pill
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Sugar Pill | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10 [6 to 17] | 8 [5 to 15] | 8 [5 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 0 | 1
  Not Hispanic | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: End-systolic Elastance
Description: end-systolic elastance (often abbreviated Ees or ESPVR) is a measure of contractility (systolic function)
Time Frame: 10 minutes after imitation of dobutamine
Measure: Mean (Inter-Quartile Range); unit: Ees in mmHg/ml/m2
Groups:
- Sugar Pill: Patients will be given a one time dose of sugar pill 30 to 90 minutes prior to catheterization.During the catheterization patients will have specialized catheter placed in the heart that measures pressure and volume simultaneously. The patients will undergo an infusion of dobutamine up to 10 micrograms per kilogram per minute to mimic exercise for up to ten minutes.
  Dobutamine: Patients will receive a dobutamine infusion during catheterization.
Arm/Group | Sildenafil | Sugar Pill
Number analyzed (Participants) | 10 | 9
Ees in mmHg/ml/m2 | 0.85 [0.01 to 1.5] | 1.8 [0.74 to 2.2]

2. Secondary Outcome: End-diastolic Pressure Volume Relationship
Description: End-diastolic pressure volume relationship (EDPVR) is a measure of diastolic (relaxation) heart function
Time Frame: 10 minutes after imitation of dobutamine
Measure: Mean (Inter-Quartile Range); unit: mmHg/ms
Arm/Group | Sildenafil | Sugar Pill
Number analyzed (Participants) | 10 | 9
mmHg/ms | 499 [367 to 899] | 953 [654 to 1482]

3. Other Pre Specified Outcome: Ventricular-arterial Coupling
Description: Ventricular-arterial coupling is a measure of efficiency of ventricular work in response to the work created by the vascular tree
Time Frame: 10 minutes after imitation of dobutamine
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | Dobutamine + Sildenafil | Dobutamine + Placebo
Number analyzed (Participants) | 10 | 10
ratio | 0.01 [-0.39 to 0.25] | 0.86 [0.26 to 1.3]

4. Other Pre Specified Outcome: Preload Augmentation
Description: Preload augmentation is a measure of how quickly the heart fills with blood during exercise
Time Frame: 10 minutes after imitation of dobutamine
Measure: Mean (Inter-Quartile Range); unit: ml/m^2
Arm/Group | Sildenafil | Sugar Pill
Number analyzed (Participants) | 10 | 9
ml/m^2 | 0.04 [0.01 to 0.08] | 0.08 [0.06 to 0.14]

ADVERSE EVENTS:
Arm/Group | Sildenafil | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=10) | Sugar Pill (N=10)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=10) | Sugar Pill (N=10)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No